CLINICAL TRIAL: NCT03430856
Title: An Open Label, Multi-center, Randomized, Parallel Group Phase II/III Clinical Study to Evaluate the Efficacy and Safety of Insulin Tregopil (IN-105) Compared With Insulin Aspart in the Treatment of Patients With Type 2 Diabetes Mellitus on Stable Dose of Metformin and Insulin Glargine
Brief Title: Comparison of Insulin Tregopil (IN-105) With Insulin Aspart in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biocon Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREGO-DM2-03-I-01
Record Dates: First submitted 2017-11-17; First posted 2018-02-13 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Oral insulin
MeSH Terms: interventions — Indium-105; Insulin Aspart

STUDY DESIGN:
Intervention Model Description: Study is conducted in two parts. Part I has 3 arms and Part 2 has 2 arms.
Masking Description: Open Label Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Insulin Tregopil (IN-105) - 45mg (Experimental): Strength of each tablet is 15mg
  Interventions: Drug: Insulin Tregopil
- Insulin Tregopil (IN-105) - 30mg (Experimental): Strength of each tablet is 15mg
  Interventions: Drug: Insulin Tregopil
- Insulin Aspart (Active Comparator): Pre-filled pen: 100 U/L
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: Insulin Tregopil — Drug: Insulin Tregopil (IN-105) Mode of Administration: To be administered orally 10 ± 2 minutes prior to each major meal (breakfast, lunch and dinner) starting at the Randomization visit.
  Other Names: IN-105
  Arms: Insulin Tregopil (IN-105) - 30mg; Insulin Tregopil (IN-105) - 45mg
Drug: Insulin Aspart — Drug: Insulin Aspart Mode of Administration: To be administered within 5 minutes prior to each major meal (breakfast, lunch and dinner) starting at the Randomization visit
  Arms: Insulin Aspart

SUMMARY:
This is an open label Phase II/III study to evaluate the efficacy and safety of test drug, Insulin Tregopil (IN-105) compared with Insulin Aspart (IAsp) in Type 2 Diabetes Mellitus patients. on stable dose of Metformin and insulin Glargine. The study will be conducted in 2 parts, Part I and Part II. The study duration will be approximately 37 weeks for Part I and for Part II of the study respectively

DETAILED DESCRIPTION:
Part I of the study is a Phase II multi-center, randomized, open label clinical study to evaluate the efficacy and safety of Insulin Tregopil (2 dose levels: 30 mg, 45 mg) compared with IAsp in the treatment of T2DM patients. Part II of the study is the Phase III, multi-center, randomized, open label clinical study to evaluate the efficacy and safety of Insulin Tregopil (30 mg or 45 mg based upon the outcome of Part I data) compared with IAsp in the treatment of T2DM patients. For Part I and Part II, the study duration will be approximately 37 weeks (3 weeks Screening, 8 weeks Run-in, 24 weeks Treatment, 2 weeks Safety follow-up). An Independent Data and Safety Monitoring Board (DSMB) will evaluate the data from Part I of the study. Part II of the study will be initiated after approval from the office of Drugs Controller General of India (DCGI) and Data Safety Monitoring Board (DSMB) recommendation based on review of data from Part I of the study. In both Part I and Part II of the study, T2DM patients with glycated hemoglobin (HbA1c) 7.5 to 10% (both inclusive), on stable dose of metformin ± oral antidiabetic drugs (OADs) ± basal insulin who are eligible for insulin glargine administration as per investigator discretion and who satisfy the selection criteria will be enrolled. The eligible patients will go through a Run-in period of 8 weeks. At the end of 8 weeks Run-in period, eligibility will be checked and patients will enter the treatment period of 24 weeks and will be allocated to 3 treatment arms (Part I) or randomized to 2 treatment arms (Part II); if found eligible for randomization. A total of 90 patients in part 1 and 268 patients in part 2 will be randomised to the treatment arms from approximately 40 centers in India.

ELIGIBILITY:
Key Inclusion Criteria

* Patients with an established diagnosis of T2DM and a duration of diabetes mellitus of at least 6 months at Screening based on criteria given below as per American Diabetes Association (ADA) 2017 guidelines: i. HbA1c ≥ 6.5% OR ii. FPG ≥ 126 mg/dL. (Fasting is defined as no caloric intake for at least 8 hours.) OR iii. 2-hour prandial glucose (PG) level of ≥ 200 mg/dL during an oral glucose tolerance test (OGTT).
* Stable dose of metformin (at least 1500 mg daily [daily dose of at least 1000 mg is permitted if intolerant to 1500 mg dose]) for a period of at least 3 months prior to Screening
* Eligible for initiation of or already receiving insulin glargine
* Hemoglobin ≥ 10.0 g/Dl
* HbA1c of 7.5% to 10.0 %
* Body mass index of 18.5 to 35.0 kg/m2

Key Exclusion Criteria

* Patients with T1DM
* Treatment with glucagon-like peptide 1 agonists within 12 weeks prior to Screening
* Ongoing treatment with OADs (eg, Thiazolidinediones) contraindicated or unapproved for combination treatment with insulin
* Presence of gastrointestinal (GI) disorders or conditions known to significantly alter the absorption of orally administered drugs or significantly alter upper GI or pancreatic function
* History of ≥2 episodes of severe hypoglycemia (as per ADA 2017) within the 6 months before Screening
* History of > 1 episode of hyperglycemic hyperosmolar coma or hospitalization for uncontrolled diabetes (eg, diabetic ketoacidosis); within the 6 months prior to Screening
* Clinically significant cardiovascular and/or cerebrovascular disease within 12 months before Screening including, but not limited to unstable angina, myocardial infarction, Class III or Class IV congestive heart failure according to the New York Heart Association criteria, valvular heart disease, cardiac arrhythmia requiring treatment, pulmonary hypertension, cardiac surgery, coronary angioplasty, stroke or transient ischemic attack.
* Patients with the following secondary complications of diabetes:

  i. Active proliferative retinopathy as confirmed by a dilated ophthalmoscopy (by the investigator, site ophthalmologist or an optometrist; as per standard site practice) within 6 months prior to Screening. ii. Renal dysfunction indicated by modification of diet in renal disease estimated glomerular filtration rate < 45 mL/min/1.73 m2 and/or diabetic nephropathy and/or clinical nephrotic syndrome at Screening. iii. History or presence of severe form of neuropathy or signs and symptoms of severe cardiac autonomic neuropathy. iv. Patients with non-traumatic amputation (at any time) or clinically significant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-12-26 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subramanian Loganathan, MD, Study Director — Biocon Research Limited
Locations (1):
- Diacon Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lebovitz HE, Fleming A, Cherrington AD, Joshi S, Athalye SN, Loganathan S, Vishweswaramurthy A, Panda J, Marwah A. Efficacy and safety of Tregopil, a novel, ultra-rapid acting oral prandial insulin analog, as part of a basal-bolus regimen in type 2 diabetes: a randomized, active-controlled phase 2/3 study. Expert Opin Pharmacother. 2022 Nov;23(16):1855-1863. doi: 10.1080/14656566.2022.2141569. Epub 2022 Nov 9. PMID 36352762

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 20 sites, which were selected for recruitment, 19 sites enrolled subjects in the run-in period, of which 15 sites later assigned subjects to randomized treatment: India:20 sites
Pre-assignment Details: The trial included an 8-week run-in period and a 24-week treatment period. During the run-in period, the subjects received insulin glargine along with metformin. In total, 143 subjects entered the run-in period, of these 52 subjects were run-in failures. Hence, 91 subjects were randomly assigned to each treatment arm.
Groups:
- Insulin Tregopil (IN-105) - 45mg: At randomization, all subjects started on 45 mg mealtime insulin Tregopil (oral) in combination with insulin glargine (basal insulin, SC, once or twice daily) and metformin (oral) in a basal-bolus regimen. Insulin Tregopil was administered (oral) 10 minutes prior to each main meal, was titrated to the 2-hour PPG target of 141-179 mg/dL according to the titration algorithm. Dose adjustments were considered once/twice weekly in the initial 4 weeks, based on the 2-hour SMPG on the previous week. Basal insulin and metformin treatment continued without changing the frequency or dose.
- Insulin Tregopil (IN-105) - 30mg: SAt randomization, all subjects started on 30 mg mealtime insulin Tregopil in combination with insulin glargine (basal insulin, SC, once or twice daily) and metformin (oral) in a basal-bolus regimen. Insulin Tregopil was administered (oral) 10 minutes prior to each main meal, was titrated to the 2-hour PPG target of 141-179 mg/dL according to the titration algorithm. Dose adjustments were considered once/twice weekly in the initial 4 weeks, based on the 2-hour SMPG on the previous week. Basal insulin and metformin treatment continued without changing the frequency or dose.
- Insulin Aspart: At randomization, all subjects started on 4 units of mealtime insulin aspart (bolus insulin) in combination with insulin glargine (basal insulin, once or twice daily) and metformin (oral) in a basal-bolus regimen. Insulin aspart was administered (sc) 0-5 minutes before each main meal, was titrated to the pre-prandial glycaemic target of 71-129 mg/dL and 2-hour PPG target of 141-179 mg/dL according to the titration algorithm. Dose adjustments were considered daily based on the pre-prandial and 2-hour SMPG on the previous week. Basal insulin and metformin treatment continued without changing the frequency or dose
Period: Overall Study
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Started | 31 | 30 | 30
Exposed | 31 | 30 | 30
Completed | 29 | 27 | 29
Not Completed | 2 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Rescue criteria | 1 | 1 | 0
Not completed — Voluntary withdrawal of consent | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all randomized subjects.
Groups:
- Insulin Tregopil (IN-105) - 30mg: At randomization, all subjects started on 30 mg mealtime insulin Tregopil in combination with insulin glargine (basal insulin, SC, once or twice daily) and metformin (oral) in a basal-bolus regimen. Insulin Tregopil was administered (oral) 10 minutes prior to each main meal, was titrated to the 2-hour PPG target of 141-179 mg/dL according to the titration algorithm. Dose adjustments were considered once/twice weekly in the initial 4 weeks, based on the 2-hour SMPG on the previous week. Basal insulin and metformin treatment continued without changing the frequency or dose.
- Total: Total of all reporting groups
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart | Total
Number analyzed (Participants) | 31 | 30 | 30 | 91
Age, Continuous [Mean (Standard Deviation); unit: Year] | 52.1 (9.49) | 50.9 (9.44) | 54.5 (8.18) | 52.5 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 14 | 43
  Male | 16 | 16 | 16 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 31 | 30 | 30 | 91
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 31 | 30 | 30 | 91
Weight [Mean (Standard Deviation); unit: kg] | 68.54 (11.559) | 68.88 (9.040) | 67.76 (9.628) | 68.39 (10.048)
Height [Mean (Standard Deviation); unit: cm] | 158.84 (7.987) | 158.76 (9.268) | 158.20 (9.321) | 158.60 (8.776)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.13 (3.866) | 27.39 (3.418) | 27.13 (3.667) | 27.22 (3.618)
Duration of T2DM [Mean (Standard Deviation); unit: years] | 8.78 (7.867) | 7.83 (7.715) | 8.12 (6.788) | 8.25 (7.404)
Glycosylated haemoglobin A1c [Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin] | 8.23 (0.577) | 8.10 (0.670) | 8.07 (0.697) | 8.13 (0.646)
OAD/Basal Insulin use at Screening Number of participants (%) [Count of Participants; unit: Participants]
  Metformin alone | 4 | 2 | 0 | 6
  Metformin + other OADs | 6 | 6 | 7 | 19
  Metformin + OADs + Basal insulin | 18 | 19 | 19 | 56
  Metformin - OADs + Basal insulin | 3 | 3 | 4 | 10
Metformin dose Number of participants (%) [Number; unit: participants]
  >=1500 mg/day | 27 | 28 | 27 | 82
  <1500 mg/day | 4 | 2 | 3 | 9
Other Abnormalities, Yes or No [Number; unit: participants]
  Yes | 8 | 6 | 3 | 17
  No | 23 | 24 | 27 | 74
Active proliferative retinopathy, Yes or No [Number; unit: participants]
  Yes | 0 | 0 | 0 | 0
  No | 31 | 30 | 30 | 91
OAD use evaluated at screening [Number; unit: participants]
  Alpha Glucosidase Inhibitors | 2 | 3 | 4 | 9
  Biguanides | 31 | 30 | 30 | 91
  Blood Glucose Lowering Drugs, Excl. Insulins | 2 | 3 | 3 | 8
  Combinations Of Oral Blood Glucose Lowering Drugs | 0 | 0 | 1 | 1
  Dipeptidyl Peptidase 4 (Dpp-4) Inhibitors | 7 | 6 | 12 | 25
  Other Blood Glucose Lowering Drugs, Excl. Insulins | 0 | 1 | 2 | 3
  Sulfonylureas | 22 | 23 | 25 | 70
  Thiazolidinediones | 2 | 2 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at 24 Weeks (Part 1)
Description: The primary endpoint is change from baseline in HbA1c after 24 weeks of randomized treatment.
Time Frame: Week 0, Week 24
Population: The analysis of this efficacy endpoint was based on the full analysis set (FAS). FAS included all randomized subjects in Part 1. The statistical evaluation of the FAS was to follow the intention-to-treat (ITT) principle and subjects contributed to the evaluation 'as randomized'.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
Percentage of glycosylated hemoglobin
  Baseline (Week 0) | 8.23 (0.577) | 8.10 (0.670) | 8.07 (0.697)
  Week 24 | 8.38 (1.139) | 8.21 (0.969) | 7.29 (0.788)
Statistical Analysis 1: Comparison: Insulin Tregopil (IN-105) - 45mg vs Insulin Aspart; Test type: Non-Inferiority — Change from baseline in HbA1c at 24 weeks of treatment, was analyzed using mixed model for repeated measures (MMRM) where all available post-baseline HbA1c measurements obtained up to Week 24 was entered as the dependent variables; visit and treatment were included as fixed factors, with Baseline HbA1c and stratification factor variables as covariates. Furthermore, the interaction terms of visit by treatment, visit by stratification factors and visit by Baseline HbA1c were included in the model; Mean Difference (Net) = 0.99, 95% CI 2-sided [0.502 to 1.470] — Insulin Tregopil 45 mg - Insulin Aspart
Statistical Analysis 2: Comparison: Insulin Tregopil (IN-105) - 30mg vs Insulin Aspart; Test type: Non-Inferiority — Non inferiority margin is 0.4%; Mean Difference (Net) = 0.89, 95% CI 2-sided [0.414 to 1.370] — Insulin Tregopil 30mg - Insulin Aspart

2. Secondary Outcome: Change From Baseline in HbA1c at Week 12 (Part 1)
Description: This secondary outcome is the change from baseline in HbA1c after 12 weeks of randomized treatment. For this endpoint baseline (Week 0) and Week 12 have been presented.
Time Frame: Week 0, Week 12
Population: This endpoint was summarized using ITT analysis set in Part I. ITT set included all randomized subjects. At Week 12, data from available participants are summarized.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
Percentage of glycosylated haemoglobin
  Baseline (Week 0) | 8.23 (0.577) | 8.10 (0.670) | 8.07 (0.697)
  Week 12: number analyzed (Participants) | 30 | 29 | 29
  Week 12 | 8.04 (0.940) | 8.01 (0.898) | 7.18 (0.810)
  Change from Baseline: number analyzed (Participants) | 30 | 29 | 29
  Change from Baseline | -0.17 (0.913) | -0.07 (0.866) | -0.88 (0.850)

3. Secondary Outcome: Participants Achieving HbA1c < 7% (Part 1)
Description: Number of participants achieving HbA1c < 7% at Week 12 and Week 24.
Time Frame: Week 12, Week 24
Population: This endpoint was summarized using intention-to-treat (ITT) analysis set. ITT set included all randomized participants. At Week 12 and Week 24, data from available participants are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
Participants
  Week 12: number analyzed (Participants) | 30 | 29 | 29
  Week 12 | 4 | 3 | 13
  Week 24: number analyzed (Participants) | 29 | 27 | 29
  Week 24 | 2 | 2 | 10

4. Secondary Outcome: Percentage of Participants With Hypoglycemia Events During 24-week Treatment Period (Part 1)
Description: A hypoglycemic episode is defined as any time a participant feels that he/she is experiencing a sign or symptom that is associated with hypoglycemia, or has blood glucose concentration of ≤ 70 milligrams/deciliter [mg/dL (3.9 millimoles/liter (mmol/L)]
Time Frame: Week 0 through Week 24
Population: This endpoint was summarized using safety analysis set in Part I. Safety analysis set included patients who were randomized and took at least 1 dose of the study drug. Patients in the safety analysis set contributed to the evaluation 'as treated'.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
Participants | 26 | 26 | 25

5. Secondary Outcome: Weight (Kgs) (Part 1)
Description: Change from Baseline in weight (kgs) to 24 weeks
Time Frame: Week 0 and Week 24
Population: This endpoint was summarized using completed participants at Week 24 and all randomised participants at Week 0 in Part I. Change from baseline was summarised using completed participants.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
Kg
  Baseline (Week 0) | 68.54 (11.559) | 68.88 (9.040) | 67.76 (9.628)
  Week24: number analyzed (Participants) | 29 | 27 | 29
  Week24 | 68.98 (11.837) | 70.15 (8.915) | 68.47 (9.761)
  Change from Baseline: number analyzed (Participants) | 29 | 27 | 29
  Change from Baseline | 0.93 (1.212) | 0.30 (1.955) | 0.66 (1.807)

6. Secondary Outcome: Lipid Profile (Part 1)
Description: Change from Baseline in lipid profile (triglycerides, low-density lipoprotein, high-density lipoprotein, and total cholesterol) to 24 weeks
Time Frame: 24 weeks
Population: This was planned for part 2 of the study. As part-2 of the study was discontinued, this is not applicable.
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Post-prandial Glucose (PPG) Excursion (Part 1)
Description: Change from Baseline in the mean 60, 90, 120 minutes PPG excursions assessed from standardized test meal at Week 24.
Time Frame: Week 0, Week 24
Population: This endpoint was summarized using the intention-to-treat (ITT) analysis set from Part I. ITT set included all randomized participants. At Week 24, data from available participants are summarized.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
mg/dL
  Week 0, 60 min | 79.5 (45.53) | 98.3 (41.94) | 74.4 (42.85)
  Week 0, 90 min | 92.4 (47.94) | 106.4 (35.39) | 90.8 (35.35)
  Week 0, 120 min | 100.9 (58.18) | 113.5 (53.45) | 93.7 (41.20)
  Week 24, 60 min: number analyzed (Participants) | 29 | 26 | 27
  Week 24, 60 min | 35.8 (44.26) | 32.7 (45.13) | 55.1 (34.57)
  Week 24, 90 min: number analyzed (Participants) | 29 | 26 | 27
  Week 24, 90 min | 53.8 (45.38) | 47.2 (44.84) | 66.3 (36.13)
  Week 24, 120 min: number analyzed (Participants) | 29 | 26 | 27
  Week 24, 120 min | 64.1 (51.87) | 50.2 (44.23) | 65.5 (34.58)

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Part 1)
Description: Includes participants who have experienced at least one treatment emergent adverse events over 24 weeks
Time Frame: 24 weeks
Population: This endpoint was summarized using Treatment Emergent Adverse Events - Safety Analysis Set (Part I).
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
Participants | 5 | 6 | 4

9. Secondary Outcome: Anti-drug Antibody Levels
Description: Incidence and change from baseline in the relative levels of anti-drug antibody levels over 24 weeks
Time Frame: 24 weeks
Population: This was planned for part 2 of the study. As part-2 of the study was discontinued, this is not applicable.
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: CGM
Description: Area under the glucose curve below 70 mg/dL derived from CGM, applicable for only part II study
Time Frame: 24 weeks
Population: This was planned for part 2 of the study. As part-2 of the study was discontinued, this is not applicable.
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 0 | 0 | 0

11. Other Pre Specified Outcome: Participants Achieving HbA1c < 7% Without Reported Clinically Significant or Severe Hypoglycemic Event Between End of Week 8 and Week 24
Description: Number of participants achieving HbA1c < 7% at Week 12 and Week 24 without reported clinically significant or severe hypoglycemic events between end of Week 8 and Week 24.
Time Frame: Week 12, Week 24
Population: This endpoint was summarized using intention-to-treat (ITT) analysis set in Part I. ITT set included all randomized participants. At Week 12 and Week 24, data from available participant are summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
Number analyzed (Participants) | 31 | 30 | 30
Participants
  Week 12: number analyzed (Participants) | 28 | 27 | 25
  Week 12 | 4 | 3 | 11
  Week 24: number analyzed (Participants) | 22 | 23 | 14
  Week 24 | 1 | 3 | 7

ADVERSE EVENTS:
Time Frame: From the date on or after first day of exposure to randomized treatment until the last day of randomized treatment, an average of 24 weeks.
Description: Safety analysis set was used for the assessment of safety including AEs. The safety analysis set included all subjects who received at least one dose of test product.
Arm/Group | Insulin Tregopil (IN-105) - 45mg | Insulin Tregopil (IN-105) - 30mg | Insulin Aspart
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/31 | 5/30 | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Tregopil (IN-105) - 45mg (N=31) | Insulin Tregopil (IN-105) - 30mg (N=30) | Insulin Aspart (N=30)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vulval laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT03430856/Prot_SAP_000.pdf